CLINICAL TRIAL: NCT03372005
Title: The Effect of Floorball on Health Parameters and Performance in Subjects With Lifestyle Diseases
Brief Title: The Effect of Floorball on Health and Performance in Subjects With Lifestyle Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Assistant professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Floorball
Record Dates: First submitted 2017-11-17; First posted 2017-12-13 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Type2 Diabetes, Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Floorball (Experimental): The subjects in this group are set to play floorball three times pr. week for 39 weeks.
  Interventions: Behavioral: Floorball
- Control (No Intervention): This group functions as a control group, that will continue the normal lifestyle throughout the study.

INTERVENTIONS:
Behavioral: Floorball — This intervention will have one week of testing before the first 12 weeks of floorball, followed by one week of testing before the last 27 week training period.
  Arms: Floorball

SUMMARY:
To investigate the effect of floorball on health and performance in subjects with either type 2 diabetes or cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Diagnosed with a cardiovascular disease (bp >140/90mmHg)
* Physical activity <2 hours pr. week.
* Not participating in any regular physical activity the last 2 years

Exclusion Criteria:

* age <18 years
* Injuries that prevent the subject from playing floorball
* Type 1 diabetics
* Alcohol >14 units pr. week.
* Pregnancy
* Participation in other scientific studies
* Abuse of illegal drugs
* other known serious diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2020-06-27 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Changes from baseline measured after 12 weeks and 39 weeks
  Long term blood sugar concentration
Blood pressure | Changes from baseline measured after 12 weeks and 39 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark